CLINICAL TRIAL: NCT04230317
Title: The Feasibility of Low Dose Chest CT for Virtual Bronchoscopy Navigation in Human Patients.
Brief Title: The Feasibility of Low Dose Chest CT for Virtual Bronchoscopy Navigation - Human Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NRF-2018R1D1A1B07046024
Record Dates: First submitted 2020-01-05; First posted 2020-01-18 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Bronchoscopy
Keywords: Computer simulation, Multislice computed tomography

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose chest CT simulation (Experimental): VBN result driven using raw data acquired with low dose CTs taken with three different protocols
  Interventions: Diagnostic Test: Chest CT
- Standard protocol chest CT simulation (Active Comparator): VBN result driven using raw data acquired with standard protocol CT
  Interventions: Diagnostic Test: Chest CT

INTERVENTIONS:
Diagnostic Test: Chest CT — Low dose CT taken with three different protocols

SUMMARY:
Advances in medical imaging technology have made it possible to detect patients with small-sized lung lesions early. Generally, invasive methods such as PCNA were used to diagnose peripheral lung nodule. However, Radial probe endobronchial ultrasonography (RP-EBUS) is widely used in the histological diagnosis of peripheral lung nodule in recent years. In order to carry out RP-EBUS, it is necessary to know the path to the lesion to access it. Conventionally, the path to the peripheral lung nodule is identified by the drawing, but recently, the path is reviewed by the virtual bronchoscopy navigation (VBN) which is reconstructed 3-dimension image using the CT data. Currently, VBN is driven by using raw data acquired using standard thin sectioned chest CT protocol, but the problem is that additional doses of radiation are exposed to patients who have initially discovered lung lesions using low dose CT. Therefore, we conduct a randomized controlled trial to verify the suitability of VBN using the raw data acquired by low dose CT.

DETAILED DESCRIPTION:
The standard thin sectioned protocol CT consists of scout, enhanced and non-enhanced image. Therefore, in this study, non-enhanced protocol CT was taken with low dose protocols with three different radiation doses to acquire raw data and drive VBN, and compared with the VBN result driven with raw data obtained with standard protocol. The primary endpoint of this study is to verify the consistency and accuracy of the VBN results driven by the raw data obtained with the low dose protocol CT.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Patients older than 18 years
   2. Competent to give informed consent
   3. Patients requiring a pathological diagnosis of pulmonary nodules using RP-EBUS.
   4. Patients who need chest CT before RP-EBUS.
2. Exclusion Criteria:

   1. Pregnancy
   2. Patients who could not receive chest CT
   3. Inability to obtain informed consent
   4. Patients unable to perform RP-EBUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Concordance rate of VBN simulation results | From CT scan to VBN drive (an average of 1 week)
  Concordance rate comparing the VBN result driven based on raw data acquired with low dose CTs taken with three different protocols compared to the VBN result driven based on raw data obtained with standard protocol CT.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Seop Eom, Study Chair — Pusan university hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim I, Lee G, Eom JS, Ahn HY, Kim A. Feasibility of low dose chest CT for virtual bronchoscopy navigation in a porcine model. Respir Res. 2019 Jul 8;20(1):142. doi: 10.1186/s12931-019-1109-8. PMID 31286968